CLINICAL TRIAL: NCT04077372
Title: A Randomized, Controlled Trial Examining the Use of The "Serious Illness Conversation Guide" (SICG) in Patients With Advanced Gastro-Intestinal Cancers
Brief Title: Assessment of a Serious Illness Conversation Guide (SICG) in Advanced Gastro-Intestinal Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-51256; VAR0179 (Other: OnCore); IRB-51256 (Other: Stanford IRB); NCI-2019-07235 (Other: NCI Trial Identifier)
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-04

CONDITIONS: Gastrointestinal Cancer; Colorectal Cancer; Pancreatic Adenocarcinoma; Gastric Cancer; Esophageal Cancer; Cholangiocarcinoma; Hepatocellular Carcinoma; Neuroendocrine Tumors; GIST, Malignant
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Cholangiocarcinoma; Carcinoma, Hepatocellular; Neuroendocrine Tumors; Gastrointestinal Stromal Tumors | interventions — Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious illness conversation guide (SICG) (Experimental): Patients have "serious illness conversation" within 3 wks of randomization and every 3 months thereafter.
  Interventions: Behavioral: Serious Illness Conversation Guide (SICG); Behavioral: Quality of Life (QOL) survey
- Conversations by treating team (Active Comparator): Patients have conversations as determined by treating team (but not using SICG tool).
  Interventions: Behavioral: Quality of Life (QOL) survey

INTERVENTIONS:
Behavioral: Serious Illness Conversation Guide (SICG) — The Serious Illness Conversation Guide (SICG) is a structured communication template designed to provide effective tool in initiating advanced care planning discussion with patients.
  Arms: Serious illness conversation guide (SICG)
Behavioral: Quality of Life (QOL) survey — Quality of life survey by questionnaire (FACT-G) given every three months

SUMMARY:
The purpose of the study is to determine whether standardized implementation of a scripted template for discussing important issues that arise near the end of life improves the care of those who have advanced cancer.

DETAILED DESCRIPTION:
Primary Objective: To determine whether the Serious Illness Conversation Guide will improve the consistency with which providers have and document conversations regarding patients' goals and priorities as they near the end of life.

Secondary Objectives: 1. To assess whether having conversations as per this model will improve the quality of care near the end of life as determined by appropriate care in concordance with their goals of care.

2. To assess whether having conversations as per this model will improve patient Quality of Life (QOL) as per a validated scale.

3. To assess in patients with concordant care whether this model will improve patient QOL as per a validated scale 4. To assess provider opinions about end-of-life conversations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer whose tumor has progressed on both FOLFOX and FOLFIRI.
* Exception: Patients with metastatic colorectal cancer whose tumors demonstrate a BRAF V600E mutation may be enrolled regardless of prior chemotherapy.
* Exception: Patients whose tumors are MSI-H must have experience progression through immunotherapy in addition to the therapies mentioned above.
* Patients with metastatic pancreatic adenocarcinoma.
* Patients with metastatic gastric or esophageal cancer whose tumor has progressed through first-line chemotherapy of any type.
* Patients with metastatic cholangiocarcinoma whose tumor has progressed through first-line chemotherapy of any type.
* Patients with metastatic hepatocellular carcinoma whose tumor has progressed through PD1 blockade.
* Patients with metastatic high-grade neuroendocrine tumor.
* A patient with a metastatic GIST that has progressed through first-line tyrosine kinase inhibitor.
* Expected life expectancy of at least one month

Exclusion Criteria:

* Any patient not meeting the above criteria
* Non-English speaking patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-10-11 (Actual)

PRIMARY OUTCOMES:
Difference in proportions of patients with documented goals of care | 1 year
  Difference in proportions of patients who have documented goals of care in medical records, assessed after death, for both arms

SECONDARY OUTCOMES:
Difference in proportions of patients with appropriate care toward end of life | 1 year
  Proportion of patients receiving appropriate care in line with their goals of care toward the end of life, by arm will be assessed.
Comparison of QOL survey measures by section | 1 year
  Comparison of survey QOL measures by section for control and intervention arms will be done by Functional Assessment of Cancer Therapy (FACT-G) , version 4 scale. It is a 28-item validated QoL questionnaire in patients receiving cancer treatment. All subscales are summed together to arrive at a total score. A higher point value is considered a better quality of life score
Overall comparison of QOL survey | 1 year
  Comparison of survey QOL measures overall for control and intervention arms will be done by Functional Assessment of Cancer Therapy (FACT-G) , version 4 scale. It is a 28-item validated QoL questionnaire in patients receiving cancer treatment. All subscales are summed together to arrive at a total score. A higher point value is considered a better quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Tyler P Johnson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT04077372/ICF_001.pdf